CLINICAL TRIAL: NCT04252612
Title: Biological Outcomes of Pramlintide in Resectable Cutaneous Squamous Cell Carcinoma: A Pilot Study
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19708
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cutaneous Squamous Cell Carcinoma
MeSH Terms: interventions — pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: Pramlintide 60 mcg twice daily (Experimental): Participants will self inject Pramlintide 60 mcg twice daily for two weeks prior to surgical resection of tumor.
  Interventions: Drug: Pramlintide
- Cohort 2: Pramlintide 60 mcg three times daily (Experimental): Participants will self inject Parmlintide 60 mcg three times daily for two weeks prior to surgical resection of tumor.
  Interventions: Drug: Pramlintide
- Cohort 3: Pramlintide 120 mcg three times daily (Experimental): Participants will self inject Parmlintide 120 mcg three times daily for two weeks prior to surgical resection of tumor.
  Interventions: Drug: Pramlintide

INTERVENTIONS:
Drug: Pramlintide — SymlinPen is a 2.7 ml; 1000 mcg/ml disposable injector pen that delivers 60 or 120 mcg doses of Pramlintide.
  Other Names: Symlin; SymlinPen

SUMMARY:
This study will treat resectable cutaneous squamous cell carcinoma patients with pramlintide for two weeks prior to surgical resection of their tumor. Pre-treatment and surgical resection specimens will then be analyzed for biological alterations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cutaneous squamous cell carcinoma. Mixed histologies (basaloid, spindle, sarcomatoid, etc.) are allowed if the pathology review favors squamous cell carcinoma as the majority component. Cancers of unknown primary sites are allowed if the clinical history and the site are highly suggestive of a skin cancer primary
* Tumor site must be amenable for surgical resection and accessible for pre-treatment biopsy
* Tumor site must be measurable by caliper measurements or by Response Evaluation Criteria in Solid Tumors (RECIST)1.1 imaging - lesions must be ≥1 cm
* Eastern Cooperative Oncology Group (ECOG) ≤2 and be medically able to undergo surgical resection
* Laboratory Requirements: Hemoglobin ≥ 8 g/dl, Platelet count ≥ 50,000/dl, Serum Creatinine ≤ 1.5 mg/dL OR Glomular Filtration Rate (GFR) ≥ 40, Serum aspartate aminotransferase (AST) and alanine transaminase (ALT) < 2.5x ULN; Total Bilirubin < 1.5x ULN (for patients with documented history of Gilbert's syndrome, total bilirubin level should be < 3.0 X ULN)
* Ability to understand and willingness to sign a written informed consent document
* Patients with child bearing potential must be willing to use barrier protection to prevent pregnancy while on study therapy and up to 30 days after the last dose of pramlintide
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Patients must be willing to comply with the protocol for the duration of the treatment including daily sub-cutaneous (SQ) injections, biopsies, scheduled visits and examinations, radiologic studies, and surgical resection

Exclusion Criteria:

* Type I diabetes: Type II diabetics (DM2) on insulin are allowed, however, for those DM2 patients that are on short acting insulin, the insulin dose should be reduced 50% and need to have regular glucose monitoring (see section 6.2.1). Type II diabetics not on insulin will not be eligible.
* Patients with known gastroparesis
* Patients with known allergic reactions to pramlintide or its ingredients
* Pregnant women and/or nursing patients will be excluded from this study because of unknown risks to fetus or nursing infants
* Any serious or uncontrolled medical disorder that could interfere with the current study as deemed by the investigating physician
* Participation in any other clinical study using an investigational agent within 21 days of starting treatment on this protocol
* No prior chemotherapy, radiation, or other tumor directed therapy within 21 days prior of starting treatment on this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Participant Compliance | at 14 days from on study date
  Patients who complete at least 75% of the injections and have not missed 2 consecutive days of treatment will be considered compliant.

SECONDARY OUTCOMES:
Number of Adverse Events | at 44 days from on study date
  Number of adverse events prior to surgery, during surgery and for 30 days after surgery that may be related to pramlintide injection.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided